CLINICAL TRIAL: NCT00830414
Title: A Pivotal Study to Evaluate the Bioequivalence of 150 mg/1 mL Medroxyprogesterone Acetate Injection in Postmenopausal Women
Brief Title: Medroxyprogesterone Acetate Injection 150 mg/1 mL in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LA486
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: medroxyprogesterone acetate
- 2 (Active Comparator): DEPO-PROVERA®
  Interventions: Drug: medroxyprogesterone acetate

INTERVENTIONS:
Drug: medroxyprogesterone acetate — IM Injection
  Arms: 1
Drug: medroxyprogesterone acetate — IM injection
  Other Names: DEPO-PROVERA®
  Arms: 2

SUMMARY:
This study compared the rates and extents of medroxyprogesterone absorption from two medroxyprogesterone acetate injection formulations following single 150 mg intramuscular (IM) injections to healthy postmenopausal women.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Screening Demographics: All volunteers selected for this study will be healthy postmenopausal women 45 years of age or older at the time of dosing. The weight range will not exceed ±20% for height and body frame as per Desirable Weights for Women - 1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and pulse, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

Screening will include a Gynecological examination (PAP smear, breast) which does not show clinically relevant findings, e.g. a cytological smear classified according to Papanicolau (PAP) higher than grade II.

The screening clinical laboratory procedures will include:

* HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
* CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
* HIV antibody, hepatitis GB surface antigen, and anti hepatitis C virus screens
* URINALYSIS: by dipstick; full microscopic examination if dipstick positive
* URINE DRUG SCREEN: amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, and opiates
* Ethyl alcohol will be measured using breath test (alcomat)
* FSH (to verify postmenopausal status)
* 17β-Estradiol (to verify postmenopausal status)
* SERUM PREGNANCY SCREEN

Is female and:

o Is postmenopausal for at least 1 year and has a serum FSH level greater than or equal to 30 mIU/mL and a serum 17β-estradiol level less than 30 pg/mL.

Exclusion Criteria

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, gynecologic or neurologic system(s) or psychiatric disease (as determined by the clinical investigators or co-investigators).
* Volunteers whose clinical laboratory test values show clinically relevant deviations from normal when confirmed on re-examination.
* Volunteers demonstrating a positive hepatitis B surface antigen screen, a positive anti HCV screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Volunteers demonstrating a positive pregnancy screen.
* Volunteers with a history of allergic response(s) to medroxyprogesterone acetate or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a history of undiagnosed vaginal bleeding.
* Volunteers with personal or immediate family (mother, sister, daughter) history of breast cancer.
* Volunteers with a history of thromboembolic disorder, thrombophlebitis, or history of anticoagulant use other than aspirin.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators or co-investigators).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 450 mL of blood within 30 days prior to dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to dosing (for hormone replacement therapy (HRT) 4 weeks prior to dosing).

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2002-04; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Horst Jurgen Heuer, M.D., Principal Investigator — AAI
Locations (1):
- AAI Deutschland GmbH & Co. KG, Neu-Ulm, Germany